CLINICAL TRIAL: NCT06892496
Title: Patient-reported Outcomes of Donor Site Healing Using Different Palatal Protection Techniques: a Randomized Controlled Clinical Trial
Brief Title: Patient-reported Outcomes of Donor Site Healing Using Different Palatal Protection Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20028832
Record Dates: First submitted 2025-03-07; First posted 2025-03-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Mucosal Erosion; Gingival Recession
Keywords: soft tissue graft; pain; wound healing
MeSH Terms: conditions — Gingival Recession; Pain | interventions — Surveys and Questionnaires; Methods; Functional Residual Capacity

STUDY DESIGN:
Intervention Model Description: The study team will assign randomly which palatal post-operative protection technique the patient will undergo by utilizing a dedicated software (Research Randomizer). The study team will then initiate the fabrication of the palatal stent in cases where VFR or 3DS groups are assigned to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vacuum-formed retainer (VFR): plastic device (Experimental): Subjects will have both dental arches scanned using an intraoral optical scanner to generate the digital model of the jaw.. A resin model will be 3D printed generating the physical model. A palatal stent will be made out of thermoforming plastic in the model using a vacuum, The stent will cover the palate and the anterior and posterior teeth, including their occlusal and buccal surfaces bilaterally, to provide retention. On the day of the surgery, at the final stage of the surgical procedure (after the graft placement and suture of the recipient site), a collagen sponge will be positioned in the palatal wound, and non-resorbable sutures will be placed above the sponge. The previously made plastic palatal stent (VFR) will be placed in position and stabilized by mechanical retention using the palate and maxillary teeth, bilaterally. The subjects will be instructed to wear the stent uninterruptedly in the first 3 days and per their preference on the 4th day and after.
  Interventions: Other: Visual Analog scale (VAS) questionnaire; Other: Vacuum-formed retainer (VFR) technique; Other: Photographs of the patient's palate; Other: Measuring graft dimensions
- 3-D printed acrylic resin stent (3DS): (Experimental): Subjects will have both dental arches scanned using an intraoral optical scanner to generate the digital model file of the patient's jaws. A palatal stent will be digitally designed. The stent will cover the palatal area to the maximum extent, respecting the limit between the hard and soft palate to avoid any discomfort or gag reflex by the subjects. At the final stage of the surgical procedure (after the graft placement and suture of the recipient site), a collagen sponge will be positioned in the palatal wound, and non-resorbable sutures will be placed above the sponge. The previously made palatal stent (3DS) will be placed in position and stabilized by mechanical retention in the palate and palatal surface of the maxillary teeth, bilaterally.
  Interventions: Other: Visual Analog scale (VAS) questionnaire; Other: 3-D printed acrylic resin stent (3DS) technique; Other: Photographs of the patient's palate; Other: Measuring graft dimensions
- Flowable resin composite stent (FRC) (Experimental): After the placement of the graft and the suture of the recipient site, a collagen sponge will be positioned in the palatal wound. Then, a layer of cyanoacrylate (PeriAcryl 90HV, GluStitch) will be placed above the sponge using a microbrush. Non-resorbable sutures will be placed covering the palatal dressing, with the suture knots facing the buccal surfaces of the maxillary posterior teeth. Finally, a layer of flowable composite will be added, covering all the wound dimensions, restricted to the wound (no extension to the adjacent teeth). Flowable composite has been shown to help reduce pain using the same principal of providing a mechanical barrier to protect the palatal wound from the oral cavity. Subjects will have both dental arches scanned using an intraoral optical scanner to generate the digital model for secondary analysis.
  Interventions: Other: Visual Analog scale (VAS) questionnaire; Other: Flowable resin composite stent (FRC) technique; Other: Photographs of the patient's palate; Other: Measuring graft dimensions

INTERVENTIONS:
Other: Visual Analog scale (VAS) questionnaire — A Visual Analog Scale (VAS) questionnaire is a type of self-report tool where respondents mark a point on a continuous line to indicate the intensity of a subjective experience, like pain, fatigue, or happiness, between two extreme anchor points (e.g., "no pain" at one end and "worst possible pain" at the other), allowing for a more nuanced response compared to a standard Likert scale; essentially, it measures the degree of a symptom along a visual continuum.
Other: Vacuum-formed retainer (VFR) technique — On the day of surgery, the stent will be positioned to cover the palate and the anterior and posterior teeth, including their occlusal and buccal surfaces bilaterally, to provide retention. Vacuum-formed retainers are a common clinical practice used after harvesting a palatal graft, in order to provide a mechanical barrier to reduce post-operative pain.
  Arms: Vacuum-formed retainer (VFR): plastic device
Other: 3-D printed acrylic resin stent (3DS) technique — On the day of surgery, the previously made palatal stent (3DS) will be placed in position and stabilized by mechanical retention in the palate and palatal surface of the maxillary teeth, bilaterally.
  Arms: 3-D printed acrylic resin stent (3DS):
Other: Flowable resin composite stent (FRC) technique — On the day of surgery, a layer of flowable composite will be added, covering all the wound dimensions, restricted to the wound (no extension to the adjacent teeth). Flowable composite has been shown to help reduce pain using the same principal of providing a mechanical barrier to protect the palatal wound from the oral cavity
  Arms: Flowable resin composite stent (FRC)
Other: Photographs of the patient's palate — At the 14-day, 30-day and 3-month follow-up visits, photographs of the patient's palate (Canon EOS 60D DSLR, Canon, USA) will be taken for healing evaluation as well as intraoral scans (TRIOS 4, 3Shape) of the palatal wound for linear and volumetric changes analysis.
Other: Measuring graft dimensions — The graft dimensions will be measured with the use of a periodontal probe and recorded on the data collection form. The professional preference in regard to technique applied and the time spent by the surgeon to adjust the stent intraorally will also be recorded in the same form.

SUMMARY:
This study has been initiated to evaluate the question, "What is the best way to protect the palate after a gum graft is removed?" The overall objective is to determine if there is a difference in PROMs of donor site healing using different palatal post-operative protection techniques.

DETAILED DESCRIPTION:
This study aims to determine if there is a difference in subject-reported outcome measures (PROMs) when different palatal post-operative protection techniques are used during healing after an autogenous soft-tissue graft is harvested from the palate for periodontal and peri-implant plastic surgery. The secondary objective is to evaluate if there is a difference in the healing of the palatal tissue via photographic and 3D linear and volumetric changes analysis after using the different protective techniques. Furthermore, the study will evaluate the time needed for fabrication and intraoral adjustment of each protective barrier and professional preference among the techniques utilized.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Healthy or Mild controlled systemic diseases with no functional limitations (ASA I or ASA II)
* Sites with 1 to 3 teeth or implants requiring soft-tissue grafting
* Minimum palatal thickness of 2 mm
* Willing to participate and sign an informed consent

Exclusion Criteria:

* Patients with systemic conditions that could impair wound healing (i.e. diabetes, immunosuppressive, chemotherapy, etc.)
* Pregnant patients
* Patients with bleeding disorders or taking anticoagulants
* Smokers
* Patients with a history of palatal graft harvesting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate postoperative pain level after autogenous gingival graft comparing 3 different palatal dressing designs | Up to 2 weeks post-operatively
  Evaluate postoperative pain level by documenting the number of pain pills taken during the initial two weeks of the healing process.
Evaluate swelling and bleeding perception after autogenous gingival graft comparing 3 different palatal dressing designs | 2 weeks, 1 month and 3 months post-operative
  Using a Visual Analog scale (VAS) questionnaire indicating the subject's perception of swelling and bleeding following the graft. The VAS is a type of self-report tool where subjects mark a point on a continuous line to indicate the intensity of a subjective experience between two extreme anchor points (e.g., "no pain" at one end and "worst possible pain" at the other), allowing for a more nuanced response compared to a standard Likert scale. Essentially, it measures the degree of a symptom along a visual continuum.
Evaluate the willingness to retreat by the subjects after autogenous gingival graft comparing 3 different palatal dressing designs | 2 weeks, 1 month and 3 months post-operative
  Using a Visual Analog scale (VAS) questionnaire indicating the subject's willingness to retreat following the graft. The VAS is a type of self-report tool where subjects mark a point on a continuous line to indicate the intensity of a subjective experience between two extreme anchor points (e.g., "no pain" at one end and "worst possible pain" at the other), allowing for a more nuanced response compared to a standard Likert scale. Essentially, it measures the degree of a symptom along a visual continuum.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Amorim Cavalcanti de Siqueira, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States